CLINICAL TRIAL: NCT00250822
Title: Single Arm, Non Randomized Phase II Trial of Gemcitabine and Oxaliplatin (GEM-OX) for Hepatocellular Carcinoma (HCC) Patients With Platelet Counts Greater Than 100,000 Per Microliter.
Brief Title: Gemcitabine and Oxaliplatin for Hepatocellular Carcinoma With Platelet Counts Greater Than 100,000 Per Microliter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0521C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-09

CONDITIONS: Liver Cancer
Keywords: Liver; hepatocellular; Gem-Ox; Cancer
MeSH Terms: conditions — Liver Neoplasms; Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine and Oxaliplatin — Dose:
  Gemcitabine 1000 mg/m2 - IV in about 60 minutes on days 1 & 15. Oxaliplatin 100 mg/m2 - IV over 2hr on days 2 & 16

SUMMARY:
To determine the primary end point response rate of the combinations of Gemcitabine and Oxaliplatin (Gem-Ox) in the treatment of hepatocellular carcinoma (HCC) in patients with platelet counts greater 100,000 per microliter in a single arme Phase II trial.

To determine the toxicity profile of this regimen To determine the effect of this treatment on patient survival, time to treatment failure, time ot progression, time to response.

DETAILED DESCRIPTION:
The treatment plan is a two-step design. Day 1 the pt will receive Gemcitabine IV and Day 2 the pt will receive Oxaliplatin IV. This treatment cycle is repeated approximately every 28 days. Subsequent treatment cycle dosages are based on toxicity diaries and lab work results. CT scans are repeated every 2 treatment cycles. Continuation in the study is dependent upon tumor response.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older, with hepatocellular carcinoma are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a ECOG performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* There must be one measurable lesion according to the RECIST criteria that should not have had prior radiation treatment.

Exclusion Criteria:

* Patients with symptomatic brain metastases that had not been adequately and definitively treated with radiation and/or surgical resection are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Life expectancy of less than 12 weeks.
* Serious, uncontrolled concurrent infection(s)
* Any prior treatment with, Gemcitabine or Oxaliplatin .
* Completion of previous chemotherapy regimen less than 4 weeks, prior to start of this study or persistence of prior treatment related toxicity.
* Treatment for other carcinomas within the last five years, except for cured non-melanoma of the skin and treated in-situ cervical cancer.
* Participation in any investigational study within 4 weeks preceding the start of the study treatment.
* Clinically significant heart disease defined as NYHA class 3 or 4 heart disease.
* Chronic debilitating diseases that the investigator feels might compromise the study Participation.
* Evidence of inadequately treated CNS metastases.
* Major surgery within 4 weeks of the s1art of the study treatment without complete recovery.
* Known or existing uncontrolled coagulopathy.
* Any of the following laboratory parameters v) Abnormal hematological values with ANC less than 1500/mm3, thrombocytopenia less than 99,000. vi) Impaired renal function with a serum creatinine of greater than 1.5 ULN vii) Serum bilirubin greater than 1.5xULN viii) Albumin less than 2.5mg/dl.
* Unwillingness to give informed consent.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response Rate ( CR + PR rate); namely, to determine response rate to the Gemcitabine and Oxaliplatin combination administered to patients with hepatocellular cancer. Furthermore, patients who achieve a response leading to tumor respectability. | Cycles will be repeated every 4 weeks until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Patt, MD, Principal Investigator — University of New Mexico
Locations (4):
- United States (4):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Lovelace Sandia Health Systems Dept of Hematology, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - St. Vincent Regional Medical Center, Santa Fe, New Mexico